CLINICAL TRIAL: NCT02410694
Title: Ixazomib in Combination With Thalidomide - Dexamethasone in Patients With Relapsed and/or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arbeitsgemeinschaft medikamentoese Tumortherapie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGMT_MM-1
Record Dates: First submitted 2015-02-09; First posted 2015-04-08 (Estimated); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — ixazomib; Thalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ixazomib-Thalidomide-Dexamethasone (Experimental): Combination therapy of:
  Ixazomib 4.0mg at days 1, 8, 15, Thalidomide 100mg at days 1 to 28 (50mg in patients aged ≥75 years), Dexamethasone 40mg (20mg in patients aged ≥75 years) at days 1, 8, 15 of a 28-day treatment cycle.
  After 8 cycles of ITD therapy, maintenance treatment with 4.0mg ixazomib (3.0mg in patients aged ≥ 75 years at first day of maintenance phase) on days 1, 8, 15 of 28-day cycles will be administered to patients with ≥ MR for a maximum period of 12 months.
  Interventions: Drug: Ixazomib; Drug: Thalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Ixazomib
Drug: Thalidomide
Drug: Dexamethasone

SUMMARY:
Overview of Study Design:

This is an open phase II, single-arm, multi-center study to evaluate progression free survival in patients receiving ixazomib in combination with thalidomide and dexamethasone (ITD) followed by an ixazomib maintenance phase of a maximum period of 12 months.

The patient population will consist of adult male and female patients with multiple myeloma (MM) with relapsed and/or refractory disease after at least one prior treatment line.

In case of enrollment patients will receive ixazomib 4.0mg at days 1, 8, 15, thalidomide 100mg at days 1 to 28 (50mg in patients aged ≥75 years), and dexamethasone 40mg (20mg in patients aged ≥75 years) at days 1, 8, 15 of a 28-day treatment cycle. The proposed number of cycles is 8. Treatment will be discontinued in case of progressive disease or in case of no response after 4 cycles (≤ SD after 4 cycles). After discontinuation of therapy an end of treatment visit (EOT) will be performed within 14 days after the last dose of the last combination treatment cycle.

After 8 cycles of ITD therapy, maintenance treatment with 4.0mg ixazomib (3.0mg in patients aged ≥ 75 years at first day of maintenance phase) on days 1, 8, 15 of 28-day cycles will be administered to patients with ≥ MR for a maximum period of 12 months. Patients who completed less than 8 cycles of ITD treatment do not qualify for maintenance phase.

Follow-up visits will be performed in 3-monthly intervals until the last patient on ixazomib maintenance therapy has concluded or discontinued the maintenance phase.

A safety analysis will be conducted after enrollment of the first 6 patients and completion of at least two cycles in every patient.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients 18 yrs or older.
2. Voluntary written consent
3. Patients in need of therapy with a diagnosis of relapsed or refractory multiple myeloma who had at least one prior treatment line
4. Patients must have measurable disease defined by at least 1 of the following criteria:

   * Serum M-protein ≥ 10g/l
   * Urine M-protein ≥ 200mg/24h
   * Serum free light chain assay: involved serum light chain ≥ 10mg/dl provided that free light chain ration is abnormal
5. Life expectancy > 3 months
6. ECOG (Eastern Cooperative Oncology Group) ≤ 2
7. • ANC ≥ 1.000/mm3 and platelet count ≥ 50.000/mm3

   * Total bilirubin ≤ 2 x ULN
   * ALT and AST ≤ 3 x ULN
   * GFR ≥ 15ml/min as calculated by cockroft-Gault equation
8. Female patients who:

   * Are older than 50 years and postmenopausal for at least 1 year before the screening visit, OR
   * Are surgically sterile, OR
   * If they are of childbearing potential, agree to practice 2 effective methods of contraception at the same time, from 4 weeks before starting study therapy through 90 days after the last dose of study drug, OR
   * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.)
   * Are informed and understand the possible consequences of the teratogenic potential of thalidomide
   * Male patients, even if surgically sterilized (i.e., status post-vasectomy), must agree to one of the following:
   * Agree to practice effective barrier contraception during the entire study treatment period and through 90 days after the last dose of study drug, OR
   * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.)
   * Are informed and understand the possible consequences of the teratogenic potential of thalidomide
9. Disease free of prior malignancies for ≥ 2 years with exception of curatively treated basal cell, squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast if they have undergone complete resection.

Exclusion Criteria:

1. lactating females or have a positive serum pregnancy test
2. Failure to have fully recovered (i.e., ≤ Grade 1 toxicity) from the reversible effects of prior chemotherapy
3. Previous treatment with ixazomib
4. Previous treatment with bortezomib or thalidomide within the last 3 months prior to baseline visit
5. Primary refractory to, or relapsing during, or within ≤ 6 weeks after end of treatment with a proteasome inhibitor and/or thalidomide
6. Previous anti-cancer treatment within the last 21 days prior to baseline visit (cycle 1 / day 1), except corticosteroid therapy (40 - 160mg dexamethasone or corticosteroid dose equivalent per month)
7. Major surgery within 14 days before enrollment
8. Radiotherapy within 14 days before enrollment. If the involved field is small, 7 days will be considered a sufficient interval between treatment and administration of the ixazomib.
9. Central nervous system involvement
10. Infection requiring systemic antibiotic therapy or other serious infection within 14 days before study enrollment
11. Evidence of current uncontrolled cardiovascular conditions
12. Systemic treatment, within 14 days before the first dose of ixazomib, with strong inhibitors of CYP1A2 (fluvoxamine, enoxacin, ciprofloxacin), strong inhibitors of CYP3A (clarithromycin, telithromycin, itraconazole, voriconazole, ketoconazole, nefazodone, posaconazole) or strong CYP3A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of Ginkgo biloba or St. John's wort
13. Ongoing or active systemic infection, active hepatitis B or C virus infection, or known human immunodeficiency virus (HIV) positive
14. Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol
15. Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent
16. Known GI disease or GI procedure that could interfere with the oral absorption or tolerance of ixazomib including difficulty swallowing
17. Diagnosed or treated for another malignancy within 2 years before study enrollment or previously diagnosed with another malignancy and have any evidence of residual disease. Patients with basal cell, squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast with are not excluded if they have undergone complete resection
18. Patient has ≥ Grade 3 peripheral neuropathy or Grade 2 with pain on clinical examination during the screening period
19. Participation in other interventional clinical trials, including those with other investigational agents not included in this trial, within 30 days of the start of this trial and throughout the duration of this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2019-03-28 (Actual); Study Completion 2019-05-02 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) | start of combination therapy to progressive disease or death due to any cause whichever occurs first, up to 4.5 years

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | best and first response since start of therapy, up to 4,5 years
Overall Survival (OS) | start of therapy to death, up to 4,5 years
Renal Response in a subgroup of patients with baseline GFR 15-30ml/min | start of therapy to best renal response, up to 4,5 years
Determination of safety by reporting of adverse events | start of therapy to end of study therapy (appr. 2 yrs)
  Reporting of adverse event as a measure of safety and tolerability
Assessment of prognostic values of risk factors at diagnosis incl. clinical assessment and cytogenetic abnormalities | screening to end of study (appr. 2 yrs)
Correlation between altered expressions of specifically selected genes and patient´s response to the treatment regimen | screening to end of study (appr. 2 yrs)

CONTACTS AND LOCATIONS:
Overall Officials: Heinz Ludwig, MD, Study Director — Wilhelminenspital Vienna
Locations (17):
- Austria (12):
  - Medizinische Universitätsklinik Graz, Klinische Abteilung für Hämatologie, Graz, Styria
  - UK Innsbruck, Universitätsklinik für Innere Medizin, Klinische Abteilung für Hämatologie und Onkologie, Innsbruck, Tyrol
  - A.ö. BK Kufstein, Abteilung für Innere Medizin, Kufstein, Tyrol
  - Ordensklinikum, KH der Barmherzigen Schwestern Linz, Interne I: Internistische Onkologie, Hämatologie und Gastroenterologie, Linz, Upper Austria
  - KH der Elisabethinen Linz, 1. Interne Abteilung, Linz, Upper Austria
  - Klinikum Wels-Grieskirchen, IV. Interne Abteilung, Wels, Upper Austria
  - LKH Feldkirch, Interne E, Feldkirch, Vorarlberg
  - Kepler Universitätsklinikum Linz, Innere Medizin 3, Zentrum für Hämatologie und medizinische Onkologie, Linz
  - Universitätsklinik der PMU Universitätsklinik für Innere Medizin III, Salzburg
  - KH der Barmherzigen Brüder Wien, Innere Medizin, Vienna
  - Med. Universität Wien, Universitätsklinik f. Innere Medizin I, Klin. Abt. f. Hämatologie u. Hämostaseologie, Vienna
  - Wilhelminenspital, Vienna
- Czechia (2):
  - Faculty Hospital Brno and Faculty of Medicine MU Brno 2nd Internal Clinic, Brno
  - Fakultní nemocnice Ostrava, Ostrava-Poruba
- Germany (3):
  - Universitätsklinikum Leipzig - AöR Selbstständige Abteilung für Hämatologie, Internistische Onkologie und Hämostaseologie, Leipzig
  - Universitätsklinikum Tübingen, Innere Medizin II, Tübingen
  - Universitätsklinikum Würzburg, Medizinische Klinik und Poliklinik II Zentrum Innere Medizin, Würzburg

REFERENCES:
- [Derived] Ludwig H, Poenisch W, Knop S, Egle A, Schreder M, Lechner D, Hajek R, Gunsilius E, Krenosz KJ, Petzer A, Weisel K, Niederwieser D, Einsele H, Willenbacher W, Melchardt T, Greil R, Zojer N. Ixazomib-Thalidomide-Dexamethasone for induction therapy followed by Ixazomib maintenance treatment in patients with relapsed/refractory multiple myeloma. Br J Cancer. 2019 Oct;121(9):751-757. doi: 10.1038/s41416-019-0581-8. Epub 2019 Sep 27. PMID 31558804